CLINICAL TRIAL: NCT00619918
Title: Nebulized Hypertonic Saline for Treatment of Viral Bronchiolitis
Brief Title: Nebulized Hypertonic Saline for Bronchiolitis
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Children's Hospital Los Angeles (Other)
Collaborators: UCSF Benioff Children's Hospital Oakland (Other); Thrasher Research Fund (Other)
Responsible Party: Principal Investigator, Susan Wu, Assistant Professor of Clinical Pediatrics, Children's Hospital Los Angeles
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CCI-06-00271
Record Dates: First submitted 2008-02-08; First posted 2008-02-21 (Estimated); Results first posted 2013-10-10 (Estimated); Last update posted 2024-11-05 (Actual); Status verified 2024-11

CONDITIONS: Bronchiolitis
Keywords: bronchiolitis; hypertonic saline
MeSH Terms: conditions — Bronchiolitis | interventions — Sodium Chloride; Saline Solution, Hypertonic; Saline Solution

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Nebulized 3% Saline (Experimental): 3% NaCl, 4 mL inhalation, up to 3 inhalations every 20 minutes in the ED, and Q8H in the inpatient setting.
  Interventions: Drug: Nebulized 3% saline
- Nebulized 0.9% Saline (Placebo Comparator): 0.9% NaCl, 4 mL inhalation, up to 3 inhalations every 20 minutes in the ED, and Q8H in the inpatient setting.
  Interventions: Drug: Nebulized 0.9% saline

INTERVENTIONS:
Drug: Nebulized 3% saline — 4 ml inhaled q8h
  Other Names: 3% saline; Hypertonic saline; NaCl 3%
  Arms: Nebulized 3% Saline
Drug: Nebulized 0.9% saline — normal saline
  Other Names: Normal saline; NS; NaCl 0.9%
  Arms: Nebulized 0.9% Saline

SUMMARY:
This study aims to examine the effect of nebulized 3% hypertonic saline in the treatment of viral bronchiolitis. The investigators hypothesize that nebulized 3% saline will decrease rate of hospital admission, decrease clinical severity scores, and decrease length of stay.

DETAILED DESCRIPTION:
Bronchiolitis is the most common viral respiratory infection in young children and infants. It is responsible for hundreds of thousands of outpatient visits and hospitalizations every year. Hypertonic saline may decrease swelling in the lung tissue, improve the patient's ability to clear secretions, and decrease nasal congestion. Hypertonic saline nebulizations have already been used effectively in patients with cystic fibrosis and in a few small trials on infants with bronchiolitis. Patients who come to the emergency department or inpatient ward of two urban free-standing pediatric hospitals in California between December and April and are diagnosed with bronchiolitis will be randomized into two groups- the control group will receive nebulized 0.9% normal saline, while the study group will receive nebulized 3% hypertonic saline. Nebulizations will be pretreated with albuterol, to prevent the theoretical risk of increased wheezing in patients with undiagnosed underlying asthma. Patients will be given up to 3 nebulizations in the emergency department, after which time the attending physician will decide whether admission to the hospital is required. Patients who are admitted will continue to receive the same nebulized treatment every 8 hours until discharged. Additional interventions such as epinephrine treatments and antibiotics can be ordered as indicated by the patient care team.

Investigators will measure symptom severity before and after treatments using the respiratory distress assessment instrument (RDAI). The investigators will compare rates of being admitted to the hospital in each group. The investigators will also compare RDAI scores, average length of stay, number of additional respiratory treatments needed, number of hours requiring oxygen, amount of IV fluid needed, and frequency of adverse effects. The investigators hypothesize that nebulized hypertonic saline will be a safe, cost-effective, and efficacious therapy which can be utilized in the outpatient setting to prevent hospital admission, as well as decrease length of stay for patients who require admission. Given the significant disease burden of viral bronchiolitis, the potential impact is substantial.

ELIGIBILITY:
Inclusion Criteria:

* clinical diagnosis of viral bronchiolitis
* between November and April

Exclusion Criteria:

* prematurity < 34 weeks
* chronic lung disease
* congenital heart disease
* history of wheezing, asthma or albuterol use
* tracheostomy status
* need for intensive care of assisted ventilation

Max Age: 24 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 447 (Actual)
Dates: Start 2008-02; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susan Wu, MD, Principal Investigator — Childrens Hospital Los Angeles/University of Southern California
Locations (2):
- United States (2):
  - Childrens Hospital Los Angeles, Los Angeles, California
  - Children's Hospital & Research Center at Oakland, Oakland, California

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wu S, Baker C, Lang ME, Schrager SM, Liley FF, Papa C, Mira V, Balkian A, Mason WH. Nebulized hypertonic saline for bronchiolitis: a randomized clinical trial. JAMA Pediatr. 2014 Jul;168(7):657-63. doi: 10.1001/jamapediatrics.2014.301. PMID 24862623

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were recruited beginning March 2008 and April 2011, only during months of bronchiolitis season (November through April). Recruitment occurred in the emergency department and general medical inpatient units at 2 urban tertiary free-standing children's hospitals in the U.S.
Pre-assignment Details: No patients were excluded after enrollment but before randomization.
Groups:
- Hypertonic Saline: 3% NaCl, 4 ml, via updraft wall nebulizer:
  * In ED: every 20 minutes up to 3 doses
  * In Inpatient: every 8 hours until discharge
- Normal Saline: 0.9% NaCl, 4 ml, via updraft wall nebulizer:
  * In ED: every 20 minutes up to 3 doses
  * In Inpatient: every 8 hours until discharge
Period: Overall Study
Arm/Group | Hypertonic Saline | Normal Saline
Started | 230 | 217
Completed | 210 | 195
Not Completed | 20 | 22
Not completed — Withdrawal by Subject | 4 | 3
Not completed — Physician Decision | 2 | 4
Not completed — Transfer to outside facility | 3 | 3
Not completed — Left before receiving first dose | 7 | 6
Not completed — ICU admission | 4 | 6

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Hypertonic Saline | Normal Saline | Total
Number analyzed (Participants) | 230 | 217 | 447
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 230 | 217 | 447
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 0.55 (0.42) | 0.53 (0.43) | 0.54 (0.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 95 | 98 | 193
  Male | 135 | 119 | 254
Region of Enrollment [Number; unit: participants]
  United States | 230 | 217 | 447

OUTCOME MEASURES:

1. Primary Outcome: Admission Rate
Description: Patients enrolled in the ED who required inpatient admission. Patients who required admission but were transferred to another facility due to lack of available beds were considered admitted for this outcome. Note, neither study site has an observation unit.
Time Frame: 1 day
Population: Analysis for this outcome only includes patients who were enrolled in the ED, and not patients enrolled in the inpatient setting.
Measure: Number; unit: participants
Arm/Group | Hypertonic Saline | Normal Saline
Number analyzed (Participants) | 196 | 183
participants
  Admitted | 55 | 76
  Discharged | 141 | 107

2. Primary Outcome: Length of Stay
Description: Length of stay defined as date of discharge minus date of admission (whole days)
Time Frame: 1 month
Population: Analysis for this outcome only includes patients who were admitted to inpatient status at the enrolling hospital and not transferred out.
Measure: Mean (Standard Deviation); unit: Days
Arm/Group | Hypertonic Saline | Normal Saline
Number analyzed (Participants) | 74 | 99
Days | 2.87 (2.00) | 2.86 (1.73)

3. Primary Outcome: Change in RDAI Score
Description: The Respiratory Distress Assessment Instrument (RDAI) is a respiratory severity score ranging from a low score of 0 to maximum score of 17. Lower scores indicate more mild symptoms; mild disease (0-6), moderate disease (7-11), and severe (12-17). A decrease in score of 2 is considered clinically significant improvement.
Time Frame: 1 Hour
Population: Excludes patients who did not receive any doses of study medication (17), patients missing pre-tx score (7), post-tx score (4), or both (1).
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Nebulized 3% Saline | Nebulized 0.9% Saline
Number analyzed (Participants) | 217 | 201
units on a scale | 1.032 (2.087) | 0.8557 (1.650)

4. Secondary Outcome: Hours of Oxygen Use
Description: Hours requiring supplemental oxygen for admitted patients.
Time Frame: 14 days
Population: Excludes patients withdrawn by investigator due to ICU admission or ineligible condition (12), withdrawn by parent (6), and missing data (3)
Measure: Mean (Standard Deviation); unit: hours
Arm/Group | Nebulized 3% Saline | Nebulized 0.9% Saline
Number analyzed (Participants) | 70 | 87
hours | 32.88 (39.99) | 31.39 (44.54)

5. Secondary Outcome: IV Fluid Use
Description: IV fluid volume administered during entire hospitalization, in mL/kg
Time Frame: 14 days
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: mL/kg
Arm/Group | Nebulized 3% Saline | Nebulized 0.9% Saline
Number analyzed (Participants) | 70 | 87
mL/kg | 51.38 (90.15) | 59.73 (107.10)

6. Secondary Outcome: Number of Participants With Supplemental Medication Use
Description: patients who received supplemental albuterol, ipratropium, or epinephrine inhaled treatment (other than pre-treatment for study med)
Time Frame: 14 days
Population: 230 patients were allocated to the 3% group; one patient allocated to the 0.9% group received 3% so was added to the 3% group for analysis, totaling 231 patients. The 0.9% group originally had 217 patients but after moving this patient to the 3% group, there are now 216 patients in the 0.9% group.
Measure: Count of Participants; unit: Participants
Arm/Group | Nebulized 3% Saline | Nebulized 0.9% Saline
Number analyzed (Participants) | 231 | 216
Participants | 39 | 39

ADVERSE EVENTS:
Time Frame: Patient enrollment through duration of hospitalization (average 3.5 days)
Description: The number of participants at risk is different from the number started because one patient randomized to the normal saline group received hypertonic saline.
Arm/Group | Hypertonic Saline | Normal Saline
All-Cause Mortality (participants affected / at risk) | 0/231 | 0/216
Serious Adverse Events (participants affected / at risk) | 0/231 | 0/216
Other Adverse Events (participants affected / at risk) | 5/231 | 8/216
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Hypertonic Saline (N=231) | Normal Saline (N=216)
ICU admission (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 6 (6) — Patients requiring admission or transfer to the PICU or NICU
Worsening cough (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 2 (2) — Parent or provider perception of worsening cough

LIMITATIONS AND CAVEATS:
* Albuterol administered before each study treatment
* Did not reach subject accrual goals
* Number of patients recruited from inpatient unit too small to analyze separately

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No